CLINICAL TRIAL: NCT07341048
Title: Characterization of Exercise Intolerance in Patients With Polycythemia Vera: Study of Potential Biological and Physiological Determinants.
Brief Title: Potential Biological and Physiological Determinants for Exercice in Patients With Polycythemia Vera
Acronym: ACTIVAQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL25_0364; 2025-A01032-47 (Other: ID-RCB)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Polycythemia; Polycythemia Vera (PV)
Keywords: Blood viscosity; polycythemia
MeSH Terms: conditions — Polycythemia; Polycythemia Vera | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Prospective, experimental, single-center, non-randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polycythemia vera (Experimental): Patients diagnosed with polycythemia vera, with confirmed presence of the JAK2 V617F mutation, who wish to resume regular daily physical activity and have been prescribed an exercise test for this purpose as part of their follow-up at Lyon Sud Hospital
  Interventions: Biological: Research samples blood viscosity and viscoelasticity:

INTERVENTIONS:
Biological: Research samples blood viscosity and viscoelasticity: — Research samples: Blood rheology: hematocrit, blood viscosity, deformability and erythrocyte aggregation, viscoelasticity
  Other Names: the level of tissue oxygenation and hemoglobin oxygenation that will be measured by near-infrared spectroscopy (NIRS).

SUMMARY:
Polycythemia vera (PV) is a rare haematological disorder characterized by an excessive production of red blood cells, associated with the somatic JAK2 V617F mutation. Clinical manifestations are varied and often include exercise intolerance but the underlying mechanisms remain poorly understood.

Physical activity is recommended in the management of chronic diseases, but it must be tailored to the physiological profile of the patient. A cardiopulmonary exercise test (CPET) is essential to ensure safety, detect possible contraindications, and assess maximal oxygen uptake (VO₂max), a key indicator of aerobic performance.

This prospective, experimental, non-randomized study will include patients with PV followed at Lyon Sud University Hospital and for which a CPET is scheduled in their routine clinical follow-up. The primary objective is to compare VO₂max between two groups of patients: moderate (<10%) versus marked (≥10%) extent of blood viscosity increase after the completion of the CPET. The main hypothesis is that a significant increase in blood viscosity during exercise (≥10%) is a major limiting factor in oxygen transport and leads to a reduced VO₂max, reflecting impaired exercise tolerance.

Secondary analyses will focus on hemorheological parameters, tissue oxygenation, and cardiorespiratory and metabolic responses. The study aims to better understand the biological and physiological determinants of exercise intolerance in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged at least 18 years and under 70.
* Patient followed for a diagnosis of Polycytemia vera (confirmed JAK2 V617F mutation) and who were prescribed a CPET because of their wish to resume regular physical activity.
* Patient affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Any known history of heart disease or chronic respiratory illness likely to affect VO₂max independently of Polycytemia vera (e.g., asthma), according to the investigator's judgment.
* Any known history of major thromboembolic complication, according to the investigator's judgment.
* Body mass index (BMI) greater than 35, according to the investigator's judgment.
* Participation in another interventional research protocol that may interfere with the present study, according to the investigator's judgment.
* Adult subject under legal protection measures (guardianship, curatorship).
* Subject currently receiving psychiatric care.
* Subject deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Blood viscosity (Centipoise) at 6 shear rates. | Measurements will be performed at baseline (pre-test), at 3 minutes post-CPET, and at 60 minutes post-CPET
  Blood viscosity will be measured using a cone-plate viscometer (Brookfield, model LVDVII+ PRO, cone CPE 40) on native hematocrit blood, at 7 different shear rates: 2.25, 4.5, 11.5, 22.5, 45, 90, and 225 s-¹, using an ascending ramp shear protocol.

SECONDARY OUTCOMES:
Rheological properties of blood: deformability and aggregation of erythrocytes | Measurements will be performed at baseline (pre-test), at 3 minutes post-CPET, and at 60 minutes post-CPET.
  Analyses will be performed on EDTA tubes. Erythrocyte deformability will be measured by ektacytometry at 9 shear stresses (0.3-30 Pa) under isotonic conditions. Maximal elongation index (EImax) and shear stress for 50% deformation (SS₁/₂) will be recorded. Aggregation/disaggregation will be assessed by syllectometry at 40% hematocrit. Parameters include aggregation index (AI) and minimal shear rate (γmin) for full disaggregation
Viscoelasticity of blood | Measurements will be performed at baseline (pre-test), at 3 minutes post-CPET, and at 60 minutes post-CPET
  Viscoelastic properties of blood will be assessed using rotational thromboelastometry (ROTEM delta) on citrated blood tubes. The following tests will be performed: NATEM, TEMACT, FIBTEM, and EXTEM. For each test, the following parameters will be measured: clotting time (CT, in seconds), clot amplitude at 5, 10, 20, and 30 minutes (A5, A10, A20, A30, in mm), alpha angle (indicating clot formation velocity, in degrees), maximum clot firmness (in mm), percentage of clot lysis at 30 minutes (LI30), as well as lysis onset time (LOT) and total lysis time (LT), both expressed in seconds
Tissue and haemoglobin oxygenation with near-infrared spectroscopy (NIRS) | Measurement will be performed during the CPET.
  Near-infrared spectroscopy (NIRS) will be performed using the Portamon MKIII system (Artinis) with a sampling rate of 100 Hz. This non-invasive technique involves placing surface electrodes on the skin over the vastus lateralis muscle, halfway between the anterior superior iliac spine and the patella. NIRS enables continuous monitoring of changes in oxyhemoglobin (HbO₂) and deoxyhemoglobin (HHb) concentrations, allowing for the calculation of the tissue oxygenation index (TOI)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine and Physical Activity. Pulmonary Function Testing. Croix Rousse Hospital., Lyon, France

IPD SHARING:
Plan to Share IPD: No